CLINICAL TRIAL: NCT02961426
Title: Open Label Phase II/III, Multicenter, Trial to Assess the Efficacy, Safety, Tolerance, and Pharmacokinetics of Sofosbuvir Plus Ravidasvir in HCV (+/- HIV) Chronically Infected Adults With no or Compensated Cirrhosis in Thailand and Malaysia
Brief Title: Strategic Transformation of the Market of HCV Treatments
Acronym: STORM-C-1
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Ministry of Health, Malaysia (Other Government); Ministry of Health, Thailand (Other Government); National Science and Technology Development Agency, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-SOF/RDV-01-HCV
Record Dates: First submitted 2016-09-07; First posted 2016-11-11 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ravidasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sofosbuvir + ravidasvir (Experimental): 12 weeks for non-cirrhotic patients, 24 weeks for cirrhotic patients
  Interventions: Drug: sofosbuvir + ravidasvir

INTERVENTIONS:
Drug: sofosbuvir + ravidasvir — combination of sofosbuvir + ravidasvir
  Other Names: ravisdasvir: PPI-668

SUMMARY:
This is a Phase II/III, multicenter, multi-country, trial to assess the efficacy, safety, tolerance and pharmacokinetics of sofosbuvir plus ravidasvir for the treatment of HCV infection.

DETAILED DESCRIPTION:
This is a Phase II/III, multicenter, multi-country trial to assess the efficacy, safety, tolerance and pharmacokinetics of SOF-RDV for the treatment of HCV infection, across genotypes 1,2,3,6, among non-cirrhotic and cirrhotic with CTP class A, interferon/ribavirin naïve or experienced, HCV mono-infected and HCV/HIV co-infected subjects.

It will also study the pharmacokinetics of RDV and, in HCV/HIV co-infected subjects, possible drug-drug interactions with antiretrovirals.

The treatment duration will be 12 weeks for subjects with no cirrhosis (Metavir F0 to F3) and 24 weeks for subjects with compensated cirrhosis (Metavir F4, CTP class A).

The study is performed in 2 stages. Stage 1 has been completed. Efficacy and safety results from Stage 1 were reviewed and approved by the independent Data and Safety Monitoring Board (DSMB) which provided the recommendation to proceed with the study stage 2. On-going stage 2 aims to supplement Stage 1 results and provide additional information on the performance of SOF-RDV in the main genotypes found in Malaysia and Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of chronic HCV infection, defined as: Positive anti-HCV antibody or detectable HCV RNA or HCV genotype at least 6 months before screening and HCV viral load ≥10^4 IU/mL at the time of screening / In subjects without documented HCV test results 6 months before screening, chronic hepatitis C infection can be assumed if risk exposures occurred > 6 months prior to screening and HCV viral load ≥10^4 IU/mL at the time of screening.
* Willing and able to provide written informed consent.
* Men and women age ≥ 18 years and < 70 years.
* Body Mass Index (BMI) of 18 to 35 kg/m2.
* Intention to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.
* Women with a negative pregnancy test at screening and baseline.
* Women of child bearing potential who accept a highly effective contraceptive method from at least 2 weeks prior to study day 1 until 1-month post-treatment. A woman is of non-child bearing potential if she (a) reached natural menopause determined retrospectively after 12 months of amenorrhea without any other obvious medical cause or (b) had procedures like bilateral tubal ligation or hysterectomy or bilateral oophorectomy.
* Subjects who are compliant in an opioid substitution maintenance program (e.g. with methadone or buprenorphine) may be included as long as there is no concern about study medications adherence and interaction or compliance to study schedules.
* Inclusion criteria related to HIV/HCV co-infected patients:

  * HIV/HCV co-infected patients receiving cART fulfilling the below criteria are eligible for the study: Antiretroviral therapy (ART) should have been initiated at least 6 months prior to screening / Patient has to have been on the same protocol-approved ARV regimen for ≥ 8 weeks prior to screening and is expected to continue the current ARV regimen through the end of study / HIV ARVs: agents allowed in this study should be administered per the prescribing information in the package insert / Screening HIV RNA < 50 copies/mL / Screening CD4 cell count ≥ 100 cells/uL
  * HIV/HCV co-infected patients not receiving cART: Screening CD4 cell count must be ≥ 500 cells/uL

Exclusion Criteria:

* Decompensated cirrhosis defined as: Evidence of advanced stage liver cirrhosis and Child-Turcotte-Pugh (CTP) Class B or C or CTP score >6) or current/past history of decompensation including ascites, variceal bleeding, spontaneous bacterial peritonitis, or hepatic encephalopathy.
* Hepatocellular carcinoma: for all patients with cirrhosis, hepatocellular carcinoma (HCC), should be excluded by liver imaging within 6 months prior to screening, and this must continue periodically as in routine HCC surveillance.
* Laboratory exclusion criteria:

  * cirrhotic subjects with albumin < 2.8 g/dL
  * direct bilirubin > 3xULN
  * AST, ALT > 10xULN
  * Low neutrophil count (≤599 cells/mm3), hemoglobin (<9.0 g/dL for male, <8.5 g/dL for female), platelets (<50000 cells/mm3 ) classified as ≥ Grade 3
* Patients with serum creatinine > 1.5 ULN or end stage renal disease
* Hepatitis B co-infection (HBsAg positive)
* Pregnancy, as documented by positive pregnancy tests at screening or baseline
* Breastfeeding
* Subjects currently receiving or unable to stop the use for at least 1 week prior to receiving the first dose of study drug any medications or herbal supplements known to be potent inhibitors or moderate inducers of cytochrome P450 (CYP) 3A4 or potent inducers of P-glycoprotein. This includes subjects who are on amiodarone or other contraindicated/excluded drugs.
* Participation in other clinical trials within 3 months.
* Any clinically significant findings or unstable condition during the screening, medical history or physical examination that, in the investigator's opinion, would compromise participation in this study as per standard guidelines and local practice. This could include patients with poorly controlled hypertension, asthma, diabetes, or other life-threatening conditions.
* Current or history of use within the preceding 6 months of immunosuppressive or immune-modulating agents. Corticosteroid used to treat any medical condition are allowed if systemic for not more than 2 weeks or if topical.
* History of solid organ or bone marrow transplantation.
* Any prior NS5A inhibitors therapy.
* Patients with significant cardiovascular conditions including:

  * myocardial infarction within the previous 6 months or
  * heart failure NYHA class III or IV
  * history of Torsade de pointes
  * Third degree heart block
  * QTcF (Fridericia) value ≥ 450 milliseconds at Baseline
  * Severe sinus bradycardia with a rate of under 50 beats per minute
  * A sinus bradycardia with third degree atrioventricular block or with Mobitz II AV block
* Use of medications associated with QT prolongation concurrently or within the 30 days prior to Screening Visit, including: macrolides, antiarrhythmic agents, azoles, fluoroquinolones, and tricyclic anti-depressants. Commonly used and essential medications for this study population like methadone and/or efavirenz is allowed as long as the QTcF value at baseline is < 450 milliseconds.
* Self-reporting active injection drug use at screening (only for stage 2).
* Exclusion criteria related to HIV/HCV co-infected patients: HIV/HCV co-infected patients not yet on stable antiretroviral therapy or for whom ART treatment initiation maybe scheduled during the study period.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response at 12 weeks post treatment completion (SVR12), as evidenced by HCV RNA level less than the lower limit of quantification | 12 weeks after the end of the study treatment
  Related objective: to assess the efficacy of sofosbuvir-ravidasvir (SOF-RDV) at 12 weeks after the end of study treatment

SECONDARY OUTCOMES:
Sustained virologic response at 4 and 24 weeks post treatment completion (SVR4 and SVR24), as evidenced by HCV RNA level less than the lower limit of quantification | 4 and 24 weeks after the end of the study treatment
  Related objective: to assess the efficacy of SOF-RDV at 4 and 24 weeks after the end of study treatment
Occurrence of on-treatment virologic failure among subjects not achieving SVR12 | 12 weeks after the end of the study treatment
  Defined as HCV RNA ≥ LLOQ at the end of the treatment period. Related objective: to assess the efficacy of SOF-RDV 12 weeks after the end of study treatment.
Occurrence of virologic breakthrough among subjects not achieving SVR12 | 12 weeks after the end of the study treatment
  Defined as either confirmed ≥ 1 log10 IU/mL increase in HCV RNA from nadir while on treatment or confirmed HCV RNA ≥ LLOQ if HCV RNA previously declined to < LLOQ while on treatment.
  Related objective: to assess the efficacy of SOF-RDV 12 weeks after the end of study treatment.
Occurrence of virologic relapse among subjects not achieving SVR12 | 12 weeks after the end of the study treatment
  Defined as HCV RNA < LLOQ at the end of the treatment period but HCV RNA ≥ LLOQ during the post-treatment period.
  Related objective: to assess the efficacy of SOF-RDV 12 weeks after the end of study treatment.
Occurrence of non-virologic failure among subjects not achieving SVR12 | 12 weeks after the end of the study treatment
  Defined as any failure that does not meet the virologic failure criteria (e.g. adverse event, lost to follow-up).
  Related objective: to assess the efficacy of SOF-RDV 12 weeks after the end of study treatment.
Occurrence of premature treatment discontinuation and occurrence of premature study discontinuation (overall and by reason for premature discontinuation) | Through study completion (up to 36 weeks for non-cirrhotic patients and up to 48 weeks for cirrhotic patients)
  Related objective: to assess the safety of SOF-RDV
Time to premature treatment discontinuation and time to premature study discontinuation | Through study completion (up to 36 weeks for non-cirrhotic patients and up to 48 weeks for cirrhotic patients)
  Related objective: to assess the safety of SOF-RDV
Occurrence of the following events: TEAE, TEAE considered to be at least possibly related to at least one of the study drugs, TEAE leading to premature treatment discontinuation, TE laboratory abnormality, grade 3/4 TEAE, TESAE and death | Through study completion (up to 36 weeks for non-cirrhotic patients and up to 48 weeks for cirrhotic patients)
  Related objective: to assess the safety of SOF-RDV. TEAE: Treatment Emergent Adverse Event TESAE: Treatment Emergent Serious Adverse Event
Time to first TEAE, time to first grade 3/4 TEAE and time to first TESAE | Through study completion (up to 36 weeks for non-cirrhotic patients and up to 48 weeks for cirrhotic patients)
  Related objective: to assess the safety of SOF-RDV. TEAE: Treatment Emergent Adverse Event TESAE: Treatment Emergent Serious Adverse Event
Maximum plasma concentration (Cmax) of ravidasvir (and sofosbuvir if needed) | Intensive PK (stage 1 only): 4 weeks after treatment initiation; Sparse PK: 4, 8 and 12 weeks after treatment initiation
  Related objective: to study the pharmacokinetics (PK) of SOF and RDV and to evaluate potential drug-drug interactions with antiretrovirals and, as needed, interactions with concomitant prescribed or non-prescribed drugs.
Baseline factors associated with SVR12 outcome | Baseline and 12 weeks after the end of the study treatment
  Related objective: to describe the subjects' demographic, clinical and biological characteristics and their relationship with SVR12.
Change in the PROQOL-HCV domain scores from treatment initiation to 12 weeks after treatment completion | 12 weeks after the end of the study treatment
  Related objective: to assess the subjects' quality of life before and after therapy.
  PROQOL-HCV: Patient Reported Outcome Quality of Life survey for HCV, questionnaire that evaluates 7 domains, each domain scores range 0 to 100, where 100 corresponds to the best quality of life.
Changes in HCV NS5A sequences from treatment initiation in subjects not achieving SVR12 | 12 weeks after the end of the study treatment
  Related objective: to evaluate the presence of viral resistance-associated variants (RAVs) to SOF-RDV in patients with virological failure 12 weeks after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Andrieux-Meyer, MD, Study Director — Drugs for Neglected Diseases; Soek-Siam Tan, MD, Principal Investigator — Selayang Hospital; Satawat Thongsawat, MD, Principal Investigator — Chiang Mai Hospital
Locations (13):
- Malaysia (9):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Department of Hepatology, Hospital Selayang, Batu Caves, Selangor
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
  - Department of Medicine/Gastroenterology, Hospital Sultanah Bahiyah, Alor Star
  - Department of Medicine/ Gastroenterology, Hospital Ampang, Ampang
  - Department of Medicine/Gastroenterology, University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan ,Pusat Penyelidikan Klinikal,Aras Bawah ,Bangunan Pengurusan,Jalan Tanah Putih, Kuantan
  - Department of Medicine/Infectious Disease, Hospital Sungai Buloh, Sungai Buloh
- Thailand (4):
  - King Chulalongkorn Memorial Hospital/HIV-NAT, Faculty of Medicine, Chulalongkorn University, Bangkok
  - Internal Medicine, Bamrasnaradura Infectious Diseases Institute, Bangkok
  - Internal Medicine unit, Medical Department, Nakornping Hospital, Chiang Mai
  - Gastroenterology unit, Department of Internal Medicine, Maharaj Nakorn Chiang Mai Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrieux-Meyer I, Tan SS, Thanprasertsuk S, Salvadori N, Menetrey C, Simon F, Cressey TR, Said HRHM, Hassan MRA, Omar H, Tee HP, Chan WK, Kumar S, Thongsawat S, Thetket K, Avihingsanon A, Khemnark S, Yerly S, Ngo-Giang-Huong N, Siva S, Swanson A, Goyal V, Bompart F, Pecoul B, Murad S. Efficacy and safety of ravidasvir plus sofosbuvir in patients with chronic hepatitis C infection without cirrhosis or with compensated cirrhosis (STORM-C-1): interim analysis of a two-stage, open-label, multicentre, single arm, phase 2/3 trial. Lancet Gastroenterol Hepatol. 2021 Jun;6(6):448-458. doi: 10.1016/S2468-1253(21)00031-5. Epub 2021 Apr 16. PMID 33865507